CLINICAL TRIAL: NCT02916238
Title: Measurement-based Care for Depression in Resource-Poor Settings
Acronym: MBC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, jessy g devieux, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIU101503WIRB20132233
Record Dates: First submitted 2016-09-24; First posted 2016-09-27 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Measurement Based Care (Experimental): Fluoxetine prescribed and dispensed beginning at 10 mg daily; side effects and symptoms monitored biweekly; dosage increased to 20 mg., then by 20 mg. increments according to protocol algorithm based on PHQ-9 score to a maximum dose of 60 mg.
  Interventions: Drug: Fluoxetine
- Enhanced Usual Care (Active Comparator): Depression symptoms monitored at 3 month interval; results from PHQ-9 available to ART clinic physicians.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine prescribed and dispensed beginning at 10 mg daily; side effects and symptoms monitored biweekly; dosage increased to 20 mg., then by 20 mg. increments according to protocol algorithm based on PHQ-9 score to a maximum dose of 60 mg.
  Other Names: Prozac
  Arms: Measurement Based Care
Behavioral: Enhanced Usual Care — Depression symptoms monitored at 3 month intervals; results from PHQ-9 available to ART clinic physicians.
  Arms: Enhanced Usual Care

SUMMARY:
Depression is often the most prevalent mental health problem among people living with HIV (PLWH) worldwide, and if not adequately treated, it may impair response to antiretroviral treatment (ART) and the ability of individuals to adhere to medications and healthy behavior. Most patients with depression receiving ART in the poorest countries of the world are left untreated because no systematic approach or expertise is available. This study adapts an evidence-based model of depression care (Measurement-Based Care - MBC) using auxiliary HIV clinic staff, and tests feasibility and assesses costs among HIV positive patients beginning ART in Port-au-Prince, Haiti.

DETAILED DESCRIPTION:
This developmental and exploratory study develops and tests a scalable model for the diagnosis and treatment of depression among HIV-infected patients initiating antiretroviral therapy (ART) in resource-poor settings. The investigators conduct a pilot test of the measurement-based care (MBC) approach to intervening, task shifting, and managing depression, which was adapted for use with auxiliary personnel who support HIV physicians in algorithm-guided antidepressant treatment. This intervention is based on the MBC approach developed by Pence, and conducted in HIV clinical sites in the US and Africa. The investigators adapted and tested an auxiliary-driven model, MBC-Aux, which is the first study of this approach with auxiliary personnel in a resource- poor country and its ART system. The study was conducted at the GHESKIO Centers in Port-au-Prince, Haiti, which is responsible for 50% of the ART population in Haiti. The investigators conducted a formative study of psychosocial factors related to depression and antidepressant medication in Aim 1, adapted the MBC depression medication and monitoring algorithm for use by auxiliary personnel at GHESKIO in Aim 2 and conducted a pre-test of procedures, and piloted the resulting MBC-Aux adaptation in Aim 3 compared to Enhanced Usual Care. The investigators also evaluated feasibility and cost. Although they are very safe medications, use of antidepressants in MBC-Aux, like use of all pharmacologic agents, incurs some measurable risk of mild, moderate and rare but severe side effects. Risks were explained to participants receiving antidepressant treatment and MBC-Aux includes systematic monitoring of participants taking these medications. This R21 developmental and exploratory study will produce the first systematic formative work of psychosocial factors related to depression in Haiti, and is the first to apply and test the MBC approach with auxiliary personnel.

ELIGIBILITY:
Inclusion Criteria:

* (1) >18, but <60 years of age; 2) able to provide informed consent; 3) documentation of HIV seropositivity; 4) ART-naïve scheduled to begin ART within 1 month; 5) total score of 10 or higher on the PHQ-9, indicating likely major depression; 6) confirmed for major depression on the MINI (Mini International Neuropsychiatric Interview);

Exclusion Criteria:

* (7) currently cognitively impaired, as determined by the MINI, since cognitive impairment may compromise the ability to comprehend and participate in the assessment and intervention; 8) bipolar disorder, psychosis, or current need for inpatient psychiatric hospitalization; 9) currently pregnant or enrolled in the GHESKIO PMTCT (Prevention of mother to child transmission) program.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Remission of Depression | 6 months
  PHQ-9 less than 5

SECONDARY OUTCOMES:
ART adherence - viral suppression | 6 months
  Improvement in Viral Load measurements
ART adherence - immune functioning | 6 months
  Improvement in CD4 measurements
Total treatment cost from the health center perspective | 6 months
  Inform a mental health intervention model for ART networks in low-and-middle income

CONTACTS AND LOCATIONS:
Overall Officials: Jessy G. Dévieux, Ph.D., Principal Investigator — Florida International University
Locations (1):
- GHESKIO Centers, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes